CLINICAL TRIAL: NCT03652662
Title: RESP-FIT: Technology-Enhanced Self-Management in COPD
Acronym: RESP-FIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00071706
Record Dates: First submitted 2018-06-26; First posted 2018-08-29 (Actual); Results first posted 2021-03-30 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This is a randomized longitudinal controlled observational study. The study will recruit 30 participants and utilize a control group experimental design with dependent pretest and posttest to derive data regarding (1) feasibility and (2) within-participant effect size of the RESP-FIT intervention in terms of satisfaction, use and adherence, technical issues and acceptability, and self-reported symptom severity (dyspnea and fatigue). When completed, 30 adults (15 in each group) will have used SAMS for 6 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RESP-FIT Intervention (Experimental): Intervention:
  IMST/EMST Training (5 breaths, 5 times a day, 5 times a week) Fitbit activity monitoring Daily symptom and training log entered into mobile application (SAMS)
  Interventions: Device: RESP-FIT
- RESP-FIT Comparator (Active Comparator): Active Comparator:
  Fitbit activity monitoring (Daily) Daily symptom and training log entered into mobile application (SAMS)
  Interventions: Behavioral: RESP-FIT Comparator

INTERVENTIONS:
Device: RESP-FIT — Inspiratory and Expiratory muscle strength training 5 times a week, plus Fitbit activity monitoring (Daily) Daily symptom and training log entered into mobile application (SAMS)
  Other Names: Combined IMST/EMST
  Arms: RESP-FIT Intervention
Behavioral: RESP-FIT Comparator — Fitbit activity monitoring (Daily) Daily symptom and training log entered into mobile application (SAMS)
  Other Names: Activity and Symptom Monitoring Only
  Arms: RESP-FIT Comparator

SUMMARY:
30 adults, aged 40 and older with mild to moderate COPD, will be recruited for this study. Participants must be willing to continually wear a FitBit activity monitor, have access to a smartphone or Wi-Fi/Data-enabled iPad, and be willing to complete respiratory muscle strength training exercises as well as reports on their smartphone at least 5 times per week for a 6-week period. Participants will be given a bluetooth inhaler device and a training app (RESP-FIT). This application will collect inhaler data and allows patients to self-report their daily symptoms. The goal of this study is to test whether use of the personalized inhaler device with the app strengthens lung function, promotes physical activity, and improves disease symptom self-management in persons with COPD.

DETAILED DESCRIPTION:
RESP-FIT. The RESP-FIT program is a 6-week respiratory muscle strength training intervention adapted from previous respiratory muscle strength training (RMST) training regimens, consisting of 1) five training days/week using combined inspiratory and expiratory muscle training, consisting of breathing in and out against a combine inspiratory and expiratory muscle strength trainer (IMST/EMST), 2) individualized, progress-based text message training reminders and prompts related to timing and intensification calibration, and 3) use of a Fitbit for remote monitoring of physical activity and hours slept at night. Similar to other muscle strength training programs, exercises are done at regular intervals during the week (5 breaths, 5 times a day, 5 days a week; the participant will receive graphical illustration of RESP-FIT training frequency and intensity achieved, and based on their training regimen, will be prompted and/or reinforced via SMS text messaging). As the use of an accelerometer or remote tracking device alone may affect physical activity, a control group will receive only the Fitbit. This study proposes to assess the feasibility and initial efficacy of RMST by obtaining estimates of variability in fatigue secondary to dyspnea, using a technologically-enhanced RESP-FIT intervention. Our overarching hypothesis is that a training regimen consisting of RMST along with technology-enhanced symptom-tracking will decrease dyspnea, dyspnea-related activity avoidance, and fatigue. Additionally, this application proposes to further develop Smartphone Airway Monitoring System (SAMS) which currently integrates EMA probe questions covering COPD symptoms and preventive care use with the new functions, use in an adult population with COPD, video captured training technique and logging of RMST training sessions. Up to thirty adults with COPD (age over 40) will complete the study and use the SAMS app for 6 weeks in the natural environment. We will evaluate the acceptability, feasibility, adherence, and performance of RESP-FIT + SAMS through quantitative methods to further optimize the app and related study procedures for the next phase of testing (i.e., large scale efficacy RCT).

ELIGIBILITY:
Inclusion Criteria:

* 40 years of age or older; and
* Able to read and write English; and
* Diagnosed with mild to moderate COPD (PFT values: FEV1/FVC <0.7 and FEV1% predicted < 50% - within the past 6 months); and
* Dyspnea score of greater than "2" on the Modified Medical Research Council (MMRC) questionnaire.

Exclusion Criteria:

* • Pregnant female or less than 1 year post-partum; or

  * Diagnosed cognitive deficit or observed lack of understanding during the informed consent process; or
  * Mobility impairment; or
  * Lack of 3g WiFi access in place of residence; or
  * Unwillingness to wear physical activity tracker daily, follow protocol, and/ or attend study visits.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2020-01-13 (Actual); Study Completion 2020-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Miller, PhD, RN, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided
As a condition of this National Institutes of Nursing Research (NINR) award, de-identified patient data will be shared by the researchers with the NINR and stored electronically on an NIH password protected secure server (https://cdrns.nih.gov/). The purpose of sharing this information is to build a NINR repository of data using Common Data Elements (CDE) for future research purposes among the general scientific community and for public health benefit.

RESULTS

PARTICIPANT FLOW:
Groups:
- RESP-FIT Intervention: Intervention:
  IMST/EMST Training (5 breaths, 5 times a day, 5 times a week) Fitbit activity monitoring Daily symptom and training log entered into mobile application (SAMS)
  RESP-FIT: Inspiratory and Expiratory muscle strength training 5 times a week, plus Fitbit activity monitoring (Daily) Daily symptom and training log entered into mobile application (SAMS)
- RESP-FIT Comparator: Active Comparator:
  Fitbit activity monitoring (Daily) Daily symptom and training log entered into mobile application (SAMS)
  RESP-FIT Comparator: Fitbit activity monitoring (Daily) Daily symptom and training log entered into mobile application (SAMS)
Period: Overall Study
Arm/Group | RESP-FIT Intervention | RESP-FIT Comparator
Started | 18 | 16
Completed | 15 | 15
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RESP-FIT Intervention | RESP-FIT Comparator | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 11 | 25
  >=65 years | 1 | 4 | 5
Age, Continuous [Mean (Full Range); unit: years] | 62 [44 to 72] | 53 [43 to 65] | 58 [43 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 5 | 6 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 15 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 11 | 11 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30
Forced Expiratory Volume by spirometry [Mean (Standard Deviation); unit: L/sec] — FEV1% is the forced expiratory volume in one second via spirometry. The unit of measure is percentage of forced expiratory in L/sec and is measured by the amount of vital capacity a person is able to expire. This was a baseline measure recorded for all participants.
  L/sec | 55.7 (17) | 55.5 (17.4) | 55.6 (17.2)

OUTCOME MEASURES:

1. Primary Outcome: Intervention Feasibility (Number of Participants Who Adhered to Treatment)
Description: Feasibility of intervention was measured by the number of participants who adhered to treatment and completed the trial (from baseline to final visit follow-up). Treatment acceptability was measured by the Mobile Application Rating Scale. The Mobile Application Rating Scale asks the participant to report the appropriateness of the app for his/her target audience ranging from little or no (1) to very high level of the acceptability measure (5).
Time Frame: through study completion, average of 6 weeks
Population: 15 participants were initially enrolled in both groups, 13 participants in the intervention group completed the trial, and 14 in the comparator group.
Measure: Count of Participants; unit: Participants
Arm/Group | RESP-FIT Intervention | RESP-FIT Comparator
Number analyzed (Participants) | 15 | 15
Participants | 13 | 14

2. Secondary Outcome: Change in Self-efficacy
Description: Change in self-efficacy (measured with the PROMIS Self-Efficacy Scale). This measures the individual's confidence in his/her ability to successfully perform specific tasks or behaviors related to one's health, with 0 being "not at all confident" to 10 being "totally confident." The PROMIS adult Self-Efficacy item banks assess self-reported current level of confidence in managing chronic conditions, including confidence in managing daily activities, managing emotions, managing medications and treatments, managing social interactions and managing symptoms.
Time Frame: baseline, 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RESP-FIT Intervention | RESP-FIT Comparator
Number analyzed (Participants) | 15 | 15
score on a scale | 6.0 (1.9) | 6.7 (2.3)

3. Secondary Outcome: Change in Fatigue
Description: Change in fatigue (measured with the PROMIS v1.0 Fatigue Scale). The PROMIS Fatigue item banks assess a range of self-reported symptoms, from mild subjective feelings of tiredness to an overwhelming, debilitating, and sustained sense of exhaustion that likely decreases one's ability to execute daily activities and function normally in family or social roles. Fatigue is divided into the experience of fatigue (frequency, duration, and intensity) and the impact of fatigue on physical, mental, and social activities. A higher PROMIS T-score represents more of the concept being measured. For negatively-worded concepts like fatigue, a T-score of 60 is one SD worse than average.
Time Frame: baseline, 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RESP-FIT Intervention | RESP-FIT Comparator
Number analyzed (Participants) | 15 | 15
score on a scale | 61.8 (8.8) | 57.8 (8.7)

4. Secondary Outcome: Dyspnea
Description: Change in difficulty breathing (measured with the PROMIS v1.0 Dyspnea). Participant can select from 5 items evaluating how shortness of breath over the past 7 days affected ability to do various activities (Getting dressed, walking stairs, household chores, or walking fast pace) ranging from "I did not do this," "no difficulty," "a little difficulty," "some difficulty," and "much difficulty." A score of 50 is the average for the general population with a standard deviation of 10 as calibration testing was performed on a large sample of the general population. The dyspnea instruments were calibrated on a sample of adults with COPD, so a score of 50 is the average for people with COPD. For the adult PROMIS Dyspnea Severity 10a short form, a raw score of 10 converts to a T-score of 48.8 with a standard error (SE) of 2.0, for an average dyspnea rating. The T-score can range from 29.7-76.7. A higher score represents more dyspnea being measured.
Time Frame: baseline, 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RESP-FIT Intervention | RESP-FIT Comparator
Number analyzed (Participants) | 15 | 15
score on a scale | 58.9 (8.8) | 55.4 (10.3)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | RESP-FIT Intervention | RESP-FIT Comparator
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 2/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RESP-FIT Intervention (N=15) | RESP-FIT Comparator (N=15)
Gastroparesis (Gastrointestinal disorders) | 0 | 1 (1) — Participant experienced gastroparesis (unrelated to study, participant was in control group)
TIA (Cardiac disorders) | 0 | 1 (1) — Participant experienced TIA (unrelated to study, participant was in control group)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-05-14): https://cdn.clinicaltrials.gov/large-docs/62/NCT03652662/Prot_SAP_000.pdf
  • Informed Consent Form (2019-05-14): https://cdn.clinicaltrials.gov/large-docs/62/NCT03652662/ICF_001.pdf